CLINICAL TRIAL: NCT00976742
Title: Impact of Common Genetic Polymorphisms on CV Disease Risk Factor Changes With Endurance Exercise Training
Brief Title: Gene - Exercise Research Study
Acronym: GERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Pittsburgh (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jim Hagberg, Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Purpose: Prevention
Other Study IDs: AG17474
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Disease Risk Factors
Keywords: plasma lipoprotein lipids; body composition; glucose tolerance; inflammation markers; insulin sensitivity; coagulation markers
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endurance Exercise Training (Experimental)
  Interventions: Behavioral: Endurance exercise training

INTERVENTIONS:
Behavioral: Endurance exercise training

SUMMARY:
The investigators hypothesize that the degree to which older generally healthy but sedentary men and women improve a number of cardiovascular (CV) disease risk factors with 6 months of highly-standardized endurance exercise training will be a function of common genetic variations in candidate genes.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* free from CV disease
* ability to undergo exercise training

Exclusion Criteria:

* previous history of CV disease

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 1998-06; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease Risk Factors | ~9 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Dept of Kinesiology, College Park, Maryland, United States

REFERENCES:
- [Result] Halverstadt A, Phares DA, Wilund KR, Goldberg AP, Hagberg JM. Endurance exercise training raises high-density lipoprotein cholesterol and lowers small low-density lipoprotein and very low-density lipoprotein independent of body fat phenotypes in older men and women. Metabolism. 2007 Apr;56(4):444-50. doi: 10.1016/j.metabol.2006.10.019. PMID 17378998